CLINICAL TRIAL: NCT06321666
Title: Response Evaluation of Cancer Therapeutics in Metastatic Breast Cancer to the Bone: A Whole Body MRI Study MILANO : RESPECT-MI
Brief Title: Response Evaluation of Cancer Therapeutics in Metastatic Breast Cancer to the Bone
Acronym: RESPECT-MI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IEO 0986
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic breast cancer; whole body magnetic resonance imaging
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WB-MRI and CT Scan (Other): CT scan (neck/thorax/abdomen/pelvis) and WB-MRI
  Interventions: Other: WB-MRI

INTERVENTIONS:
Other: WB-MRI — All patients will undergo a CT scan (neck/thorax/abdomen/pelvis) and a WB-MRI

SUMMARY:
This is a non randomized, single arm study, where each patient will undergo imaging with Computed Tomography (CT) and Whole-body magnetic resonance imaging (WB-MRI) at different timepoint. The primary endpoint is time to progression as documented by CT or WB-MRI.

DETAILED DESCRIPTION:
This is a monocentric study. All patients will undergo assessments by CT and WB-MRI at all time points.

* A baseline bone scan or Fluorodeoxyglucose-Position Emission Tomography (FDG-PET) will be performed.
* CT scans and WB--MRI are performed every 12 weeks until week 96, and then every 24 weeks until disease progression is evident (as defined in section 7.1.3).
* At the point of disease progression, a repeat bone scan or FDG-PET/CT will be obtained in addition to the CT and WB-MRI. Participation in the trials ends at the point of disease progression.

Patients will be reviewed in outpatient clinic:

* At baseline
* Every 12 weeks until week 96, with the results of their recent scans.
* As with the imaging, the trial visits will change to every 24 weeks after the week 96 visit.

At the week 12 and week 36 visits, the patients will undergo a clinical examination and perform a pain thermometer score and Patient Imaging Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of breast cancer
* Single or multiple bone metastases (additional extraosseous or non-bony metastatic disease permitted)
* Due to start a new line of either hormone therapy or chemotherapy (use of bisphosphonates / denosumab or targeted agents e.g. trastuzumab in addition to hormone therapy / chemotherapy permitted)
* Aged 18 and over
* Life expectancy of over 6 months
* No current active malignancy other than breast cancer

Exclusion Criteria:

* Radical treatment to sole site of metastatic disease e.g. Cyberknife to solitary bone metastasis
* Absolute contraindication to MRI studies, CT scans, bone scans or FDG-PET/CT
* Pregnancy
* Psychological, familial, sociological or geographical conditions that would hamper compliance with the study protocol; such conditions should be discussed with the patient as part of the informed consent process.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2019-09-12 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of disease progression in bone metastasis identified by WB-MRI prior to CT scan | 36 months
  Number of patients where disease progression in bone metastases were identified using WB-MRI prior to identification by CT scan

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Petralia, MD, Principal Investigator — European Institute of Oncology
Locations (1):
- IEO Istituto Europeo di Oncologia, Milan, Italy